CLINICAL TRIAL: NCT05770154
Title: Ankle Isokinetic Strength and Balance Assessment in Diabetic Patients With and Without Peripheral Neuropathy at Different Angular Velocities
Brief Title: Isokinetic Strength and Balance Assessment in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Other Study IDs: isokinetic in diabetic
Record Dates: First submitted 2023-02-15; First posted 2023-03-15 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Diabetes
Keywords: diabetes,; diabetic polyneuropathy; isokinetic; muscle strength; dynamic balance
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic polyneuropathy (DPN) is a type of nerve damage that can occur in diabetics. It can cause weakness and a loss of sensation, particularly in the legs and feet. This can have an impact on muscle strength and balance, making walking more difficult and increasing the risk of falling. Evaluating ankle muscular strength and balance using quantitative and standardised tools is critical for patients with and without DPN as well as determining how much DPN affects ankle muscle strength and balance.

DETAILED DESCRIPTION:
Diabetic Peripheral Neuropathy (DPN) can affect ankle muscle strength and increase the risk of falling. This occurs due to nerve damage that impairs muscle function and reduces sensitivity in the feet, leading to difficulty maintaining balance and coordination. Risk factors for DPN-related falls include poor glycemic control, the duration of diabetes, age, and other comorbidities such as peripheral vascular disease. It is important for individuals with diabetes to regularly monitor and manage their DPN to prevent falls and maintain overall health. So, conducting this study to measure ankle muscle strength through isokinetic testing and dynamic balance through the Biodex balance system will help researchers quantify the extent of DPN's impact on these aspects. This study can provide a valuable predictor and assessment tool for determining the severity of neuropathy in diabetic patients. The results of this study could also help identify those at a higher risk for falls and diabetic foot complications. This information can aid healthcare providers in developing tailored interventions to improve muscle strength and balance and reduce the risk of falls in individuals with diabetes and DPN.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 40 to 55 years for both gender.
2. Patients with diabetes for more than 5 years.
3. Diabetic polyneuropathy was diagnosed by a neurologist.
4. Their BMI from 18 to 24.9 kg/m2.
5. The study population must be willing to participate in the study.

Exclusion Criteria:

1. Patients with marked deformities of the lower limbs, foot ulcers and Charcot foot.
2. .Patients with any other neurological or orthopedic diseases that may affect balance.
3. Patients with marked weakness or drop foot.
4. Patients with amputation, mental deficits, liver or renal diseases.
5. patients who had a previous surgical history (within 6 months) were also excluded prior to the baseline assessment

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: diabetic patient
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Peak torque | Through study completion, an average of 6 months.
  Isokinetic dynamometer will be used for measuring ankle dorsi and planter flexors peak torque at different angular velocities.

SECONDARY OUTCOMES:
Power | Through study completion, an average of 6 months.
  Isokinetic dynamometer will be used for measuring ankle dorsi and planter flexors power at different angular velocities.
Work | Through study completion, an average of 6 months.
  Isokinetic dynamometer will be used for measuring ankle dorsi and planter flexors work at different angular velocities
Dynamic balance | Through study completion, an average of 6 months.
  Biodex balance system will be used to assess dynamic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Elimy, phD, Principal Investigator — Cairo University; Khaled T Ahmed, Ass. prof, Principal Investigator — Misr University for Science and Technology; Wafaa A Abd Allah, phD, Principal Investigator — Misr University for Science and Technology; Mohamed F Abdel-lateef, phD, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Doaa Ayoub Elimy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Study protocol